CLINICAL TRIAL: NCT00623259
Title: Phase I Vaccination Study Testing the Safety and Reactogenicity of a Recombinant MVA HIV Multiantigen Vaccine (MVA-mBN120B) in HIV-infected Subjects With CD4 Count > 350/µL
Brief Title: Phase I Safety Study of a Recombinant MVA HIV Multiantigen Vaccine in HIV-infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Responsible Party: Monika Fluer, Bavarian Nordic
Purpose: Diagnostic
Other Study IDs: HIV-MAG-001
Record Dates: First submitted 2008-02-19; First posted 2008-02-26 (Estimated); Last update posted 2010-05-20 (Estimated); Status verified 2010-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: MVA-mBN120B

INTERVENTIONS:
Biological: MVA-mBN120B

SUMMARY:
Monocentric study to assess the safety and immunogenicity of the recombinant MVA-HIV multiantigen vaccine MVA-mBN120B in HIV-infected subjects. 15 subjects will receive immunizations at day 0, after 4 and 12 weeks at a dose of 2E8 TCID50 MVA-mBN120B. The vaccine will be administered subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged between 18 to 55 years.
* HIV-1 infection documented by either plasma HIV-1 RT-PCR or bDNA assay at any time prior to study entry.
* Stable on HAART with regard to immunologic and clinical parameters for at least 6 consecutive months prior to study entry (substitutions of one drug for another in the same class due to reasons other than virologic failure are allowed).
* Plasma HIV RNA level < 50 copies/ml for at least 6 months prior to study entry; single blips of up to 400 HIV-1 RNA copies/ml are acceptable if they resolve spontaneously without a change in HAART.
* Plasma HIV-1 RNA levels of < 50 copies/ml at study entry.
* Women with childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours prior to immunization.
* Women of childbearing potential must have used an acceptable method of contraception for 30 days prior to the first immunization, must agree to use an acceptable method of contraception during the study, and must not become pregnant for at least 28 days after the last immunization. A woman is considered of childbearing potential unless post-menopausal or surgically sterilized. (Acceptable contraception methods are restricted to abstinence, barrier contraceptives, intrauterine contraceptive devices or licensed hormonal products.)
* CD4 cells ≥ 350/µl (two determinations, of which one must be done during the screening and the other must be done within 3 months before study entry)
* CD4 nadir > 150/µl.
* Troponin I within normal institutional limits.
* White blood cells ≥ 2500/mm3 and < = 11,000/ mm3.
* Negative urine glucose by dipstick or urinalysis at screening.
* Haemoglobin ≥ 9.0g/dL.
* Platelets ≥ 100,000/mm3
* Adequate renal function defined as:

  1. Calculated Creatinine clearance (CrCl) > 50 mL/min as estimated by the Cockroft-Gault equation.
  2. Urine protein < = 100 mg/dL or none or trace proteinuria (by urinalysis or dip stick (< = 2+ proteinuria)).
* Adequate hepatic function defined as:

  1. Total bilirubin < = 2 x ULN unless elevation is explained by antiviral therapy and in the absence of other evidence of significant liver disease (healthy subjects without clinical disease with Gilbert's Syndrome can be included).
  2. AST (SGOT), ALT (SGPT) and alkaline phosphatase < = 3 x ULN without clinically significant findings.
* Electrocardiogram (ECG) without abnormal findings (e.g. any kind of atrioventricular or intraventricular conditions or blocks such as complete left or right bundle branch block, AV-node block, QTc or PR prolongation, premature atrial contractions or other atrial arrhythmia, sustained ventricular arrhythmia, two premature ventricular contractions (PVC) in a row, ST elevation consistent with ischemia).
* Negative test for hepatitis B surface Antigen (HBsAg) and hepatitis C antibody (HCV Ab).
* Free of obvious health problems as established by medical history and physical examination before entering into the study.
* Signed informed consent form of the subject after information of the risks and benefits of the study in a language the subject clearly understands, and before any study specific procedure.
* Availability for follow-up for the planned duration of the study.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Uncontrolled serious infection i.e. not responding to antimicrobial therapy.
* History of any serious medical condition, which in the opinion of the investigator would compromise the safety of the subject.
* History of suspected or active autoimmune disease. Persons with vitiligo or thyroid disease taking thyroid replacement therapy are not excluded.
* History of chronic alcohol abuse (40g / day for at least 6 months) and/or intravenous drug abuse (within the past 6 months).
* History of malignancy, other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure. Subjects with history of skin cancer at the vaccination site are excluded.
* Manifestation of clinically significant and severe haematological, pulmonary, central nervous, cardiovascular or gastrointestinal disorder.
* Clinically significant mental disorder not adequately controlled by medical treatment.
* Any condition which might interfere with study objectives or would limit the subject's ability to complete the study or to be compliant in the opinion of the investigator.
* History of coronary heart disease, myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure, or any other heart condition under the care of a doctor.
* History of an immediate family member (father, mother, brother, or sister) who died due to ischemic heart disease before age 50 years.
* Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool. (http://hin.nhlbi.nih.gov/atpiii/calculator.asp?usertype=prof) NOTE: This criterion applies only to volunteers 20 years of age and older.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Known allergy to egg or aminoglycoside (gentamicin).
* History of anaphylaxis or severe allergic reaction.
* Having received any vaccinations or planned vaccinations with a live vaccine within 30 days prior or after study vaccination.
* Having received any vaccinations or planned vaccinations with a killed vaccine within14 days prior or after study vaccination.
* Chronic administration (defined as more than 14 days) of systemic immuno-suppressant drugs during a period starting from six months prior to administration of the vaccine and ending at study conclusion. (Corticosteroid nasal sprays are permissible. Persons who have used topical and inhaled steroids can be enrolled after their therapy is completed).
* Post organ transplant subjects whether or not receiving chronic immunosuppressive therapy.
* Any continuous therapy that may influence CD4 counts other than antiretroviral therapy.
* Administration or planned administration of immunoglobulins and/or any blood products during a period starting from 3 months prior to administration of the vaccine and ending at study conclusion.
* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days or 7 half-lives (whichever is longer) preceding the first dose of the study vaccine, or planned administration of such a drug during the study period.
* Previous participation in another HIV vaccination study.
* Previous participation in any MVA vaccination study during the last 5 years.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States